CLINICAL TRIAL: NCT05993806
Title: A Randomized, Open-label, Single-dose, Two-sequence, Two-period, Cross-over Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of L04TD3 and L04RD1 in Healthy Adult Volunteers
Brief Title: A Bioequivalence Study of L04TD3 Compared to Administration of L04RD1 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-L04-103
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (L04RD1 -> L04TD3) (Experimental): Administration of 1 tablet of L04RD1, and taking 7-day wash-out period, and then administration of 1 tablet of L04TD3
  Interventions: Drug: L04RD1; Drug: L04TD3
- B (L04TD3 -> L04RD1) (Experimental): Administration of 1 tablet of L04TD3, and taking 7-day wash-out period, and then administration of 1 tablet of L04RD1
  Interventions: Drug: L04RD1; Drug: L04TD3

INTERVENTIONS:
Drug: L04RD1 — 1 tablet of L04RD1
Drug: L04TD3 — 1 tablet of L04TD3

SUMMARY:
This is a randomized, open, single-dose, crossover-design, phase 1, singlecenter study to evaluate bioequivalence after administration of L04RD1 or administration of L04TD3 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A subject aged 19 to less than 65 years at the time of the screening visit
* A subject with a body weight of 55kg or higher and a body mass index (BMI) of 18.0 kg/m2 to 29.9 kg/m2, inclusive
* A subject considered appropriate to participate in the study according to the results of lab tests such as the hematological test, blood chemistry test, serum test, urinalysis, etc. and ECG set and conducted by the principal investigator (or a delegated study physician) according to the characteristics of the investigational product
* A subject who agreed to exclude the possibility of pregnancy by having themselves, their spouses, or partners use medically appropriate contraceptive methods and not to provide sperm or egg from the first dose to 7 days after the last dose of IP administration
* A subject who voluntarily signed the informed consent form after listening to and understanding sufficient explanation on the purpose, content of this clinical study, the characteristics of the investigational product, expected adverse events, etc.

Exclusion Criteria:

* A subject who has clinically significant diseases in the digestive system, cardiovascular system, endocrine system, respiratory system, blood and tumor, infectious disease, kidney and genitourinary system, mental and nervous system, musculoskeletal system, immune system, otolaryngeal system, skin system, and ophthalmic system or has had the diseases
* A subject who had gastrointestinal surgery (excluding simple appendectomy or hernia surgery) which may affect the absorption of drugs or have gastrointestinal diseases
* A subject who took drugs that induce and inhibit drug metabolizing enzymes such as barbiturates within one month from the first administration date or drugs that might affect this clinical study within 10 days from the first administration date (subjects may participate depending on the pharmacodynamics and pharmacokinetics such as the interactions with the investigational product, half-life, etc.)
* A subject who participated in another clinical study or bioequivalence study where they were administered the investigational product within 6 months prior to the first dose of the investigational drug
* A subject considered by the principal investigator (or a delegated study physician) as inappropriate to participate in this clinical study due to reasons other than the above inclusion and exclusion criteria

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
AUCt | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
Cmax | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours

SECONDARY OUTCOMES:
AUCinf (Area under the plasma concentration-time curve from time 0 to infinity) | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
Tmax (Time of peak plasma concentration) | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
AUCt/AUCinf | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
t1/2 (Half-life) | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours
CL/F | Pre-dose(0), 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 34.00, and 48.00 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H plus Yangji Hospital, Seoul, South Korea